CLINICAL TRIAL: NCT02435225
Title: Brain Connectivity and Mindfulness Training in Youth With Bipolar Disorder NOS
Brief Title: Brain Connectivity and Mindfulness Training in Youth With Bipolar Disorder Not Otherwise Specified (NOS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in goals of PI
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MH10126001; NCT02095483 (obsolete NCT alias)
Record Dates: First submitted 2013-08-07; First posted 2015-05-06 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Bipolar Disorder, NOS
MeSH Terms: conditions — Bipolar Disorder | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mindfulness group (Experimental): Participation in a 12 week mindfulness therapy group.
  Interventions: Behavioral: Mindfulness Based Stress Reduction for Teens Group

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction for Teens Group — A 12-Week weekly group intervention to train adolescents in mindfulness practice

SUMMARY:
The investigators propose to study 30 adolescents with bipolar disorder, not otherwise specified (BD NOS) and a family history of Bipolar I Disorder (BD) at baseline with rs-fMRI (functional magnetic resonance imaging) and functional connectivity (FC) analyses and compare data with previously acquired rs-fMRI and FC data from 20 age- and gender-matched healthy controls (HC). Subjects will then undergo a 12-week Mindfulness based stress reduction- teen (MBSR-T) intervention and be reassessed and rescanned. The intervention and scanning will take place in groups of 6-8 subjects/group/year over the 4 years. This proposal will be a natural progression of past research, while extending the investigators' expertise to include advanced FC analyses and mindfulness based interventions in youth with mood dysregulation. The investigators will also integrate trainees into the imaging and therapy components of this study, furthering our mission of mentoring the next generation of innovative researchers who will push the field forward.

ELIGIBILITY:
Inclusion Criteria:

* Ages 13-17
* Diagnosed with BD-NOS
* First or second degree relative diagnosed with bipolar I or II

Exclusion Criteria:

* Not English speaking
* For those who are to participate in the MRI scan, having any metal in the body or movement disorders will be an exclusionary factor

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Dorsal Medial Network functional connectivity | 12 weeks
  (1) Use ICA to compare DMN in subjects with BD NOS to healthy controls (HC)
Functional connectivity of sgACC with thalamus, VMPFC, and amygdala | 12 weeks
  (2) Investigate level of FC of the sgACC with thalamus, VMPFC, amygdala, and FC of pCing with amygdala/hippocampus, comparing subjects to HC.

SECONDARY OUTCOMES:
Degree of Mindfulness | 12 weeks
  Will use measures of self report to determine amount and quality of mindfulness practice and degree of daily mindfulness achieved

CONTACTS AND LOCATIONS:
Overall Officials: Kiki D Chang, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States